CLINICAL TRIAL: NCT00446264
Title: Sequential Islet Transplantation With Steroid Free Immunosuppression for Type 1 Diabetes
Brief Title: Islet Allotransplantation With Steroid Free Immunosuppression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 01/48; PHRC (Other: 2001/1939); AFSSAPS 030209 (Other: AFSSAPS)
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Results first posted 2010-05-12 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2009-02

CONDITIONS: Type 1 Diabetes; Hypoglycemia; Metabolic Diseases
Keywords: diabetes; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Metabolic Diseases; Diabetes Mellitus | interventions — Islets of Langerhans Transplantation; Tacrolimus; Sirolimus; Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- islet transplantation (Experimental): Each participant received up to three sequential fresh islet infusions within three months.
  Interventions: Procedure: islet transplantation; Drug: daclizumab - sirolimus - tacrolimus

INTERVENTIONS:
Procedure: islet transplantation — Islet transplantation consisted of up to three sequential fresh islet infusions within three months. Access to the portal vein was gained under general anesthesia by percutaneous catheterisation of a peripheral portal branch under ultrasound guidance or by surgical catheterisation of a small mesenteric vein.
  Other Names: surgical catheterisation; percutaneous catheterisation
Drug: daclizumab - sirolimus - tacrolimus — Immunosuppressive consisted of Tacrolimus, target through level at 3-6 ng/ml, Sirolimus, target through level at 12-15 ng/ml for three months and at 7-10 ng/ml thereafter. A five-dose induction course of Daclizumab 1mg/Kg was administered biweekly beginning one hour prior to the first infusion
  Other Names: Prograf; Rapamune; Zenapax

SUMMARY:
The restoration of endogenous insulin secretion carries significant hopes for shifting the paradigm of life long exogenous insulin therapy in selected groups of patients with type 1 diabetes(T1D). After decades of frustrating clinical attempts, the Edmonton group set up in 2000 new standards for islet transplantation in patients with brittle T1D by achieving insulin independence in 80 percent of patients. These seminal results have however proved much more difficult to duplicate than initially expected.

This single center phase 2 clinical trial, duplicating the Edmonton protocol, is designed for confirming the consistent short term efficacy and safety of sequential islet allotransplantation with steroid free immunosuppression in patients with severe T1D.

DETAILED DESCRIPTION:
The short term effectiveness of islet transplantation for alleviating hypoglycemia and controlling glucose homeostasis while limiting or even avoiding the nedd for exogenous insulin has been established despite protocol modifications in donor selection, islet preparation or recipient treatment, insulin independence with adequate metabolic control was however rarely prolonged beyond two years. The most frequently proposed explanations include chronic allogenic rejection, recurrence of autoimmunity and beta cell toxicity from administered immunosuppressive drugs.

Fourteen patients were enrolled in this single center phase 2 trial initiated in 2003. Eligible patients were males or females between 18 and 65 years of age, with type 1 diabeted documented for more than 5 years, arginine stimulated C-peptide lower than 0.2ng/ml, and hypoglycemia awareness or documented metabolic lability. Exclusion criteria included body mass index greater than 28Kg/m2, unstable arteriopathy or heart disease, active infection, previous transplantation, insulin daily requirements above 1.2 UI/kg, creatinin clearance below 60 ml/mn/m2 or urinary albumin excretion above 300 mg/day, malignancy, smoking, desire for pregnancy, psychiatric disorders and lack of compliance. The study primary efficacy endpoint was graft survival defined as insulin independence and HbA1c<6.5%. Secondary outcomes were graft function and metabolic control.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes documented for more than 5 years
* arginine stimulated C-peptide lower than 0.2 ng/mL
* one of the following:hypoglycemia unawareness OR metabolic lability documented by one or more severe hypoglycemias or two or more hospital admissions for ketoacidosis within the previous year.

Exclusion Criteria:

* body mass index greater than 28 kg/m2
* non stable arteriopathy or heart disease
* active infection
* previous transplantation
* hyperimmunization
* insulin daily needs above 1.2 U/Kg
* creatinine clearance below 60 ml/mn or urinary albumin excretion above 300 mg/d
* malignancy
* smoking
* desire for pregnancy
* psychiatric disorders
* lack of compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-05; Primary Completion 2007-10 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Pattou, MD, Principal Investigator — University Hospital, Lille; Marie-Christine Vantyghem, MD PhD, Principal Investigator — University Hospital, Lille; Julie Kerr-Conte, PhD, Principal Investigator — Université de Lille 2
Locations (1):
- University Hospital of Lille, Lille, France

REFERENCES:
- [Derived] Vantyghem MC, Chetboun M, Gmyr V, Jannin A, Espiard S, Le Mapihan K, Raverdy V, Delalleau N, Machuron F, Hubert T, Frimat M, Van Belle E, Hazzan M, Pigny P, Noel C, Caiazzo R, Kerr-Conte J, Pattou F; Members of the Spanish Back Pain Research Network Task Force for the Improvement of Inter-Disciplinary Management of Spinal Metastasis. Ten-Year Outcome of Islet Alone or Islet After Kidney Transplantation in Type 1 Diabetes: A Prospective Parallel-Arm Cohort Study. Diabetes Care. 2019 Nov;42(11):2042-2049. doi: 10.2337/dc19-0401. PMID 31615852
- [Derived] Benomar K, Chetboun M, Espiard S, Jannin A, Le Mapihan K, Gmyr V, Caiazzo R, Torres F, Raverdy V, Bonner C, D'Herbomez M, Pigny P, Noel C, Kerr-Conte J, Pattou F, Vantyghem MC. Purity of islet preparations and 5-year metabolic outcome of allogenic islet transplantation. Am J Transplant. 2018 Apr;18(4):945-951. doi: 10.1111/ajt.14514. Epub 2017 Nov 11. PMID 28941330
- [Derived] Caiazzo R, Vantyghem MC, Raverdi V, Bonner C, Gmyr V, Defrance F, Leroy C, Sergent G, Hubert T, Ernst O, Noel C, Kerr-Conte J, Pattou F. Impact of Procedure-Related Complications on Long-term Islet Transplantation Outcome. Transplantation. 2015 May;99(5):979-84. doi: 10.1097/TP.0000000000000458. PMID 25393157
- [Derived] Vantyghem MC, Raverdy V, Balavoine AS, Defrance F, Caiazzo R, Arnalsteen L, Gmyr V, Hazzan M, Noel C, Kerr-Conte J, Pattou F. Continuous glucose monitoring after islet transplantation in type 1 diabetes: an excellent graft function (beta-score greater than 7) Is required to abrogate hyperglycemia, whereas a minimal function is necessary to suppress severe hypoglycemia (beta-score greater than 3). J Clin Endocrinol Metab. 2012 Nov;97(11):E2078-83. doi: 10.1210/jc.2012-2115. Epub 2012 Sep 20. PMID 22996144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 2003-2006 University Lille Hospital
Groups:
- Single Arm Group: Islet Allotransplantation Group
Period: Overall Study
Arm/Group | Single Arm Group
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Group
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants] — 18-65
  Participants
    <=18 years | 0
    Between 18 and 65 years | 14
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Region of Enrollment [Number; unit: participants]
  France | 14

OUTCOME MEASURES:

1. Primary Outcome: Composite Criteria: Insulin Independence and Glycosylated Hemoglobin (HbA1c) Under 6.5% at One Year
Description: The percentage of insulin independents subjects with an HbA1c less than 6.5% at one year after last transplant
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Percentage of patients
Arm/Group | Single Arm Group
Number analyzed (Participants) | 14
Percentage of patients | 71 (29)

2. Secondary Outcome: Hypoglycemic Events
Description: Percentage of subjects free of severe hypoglycemic events from day 0 to day 365 with the day of transplant designated day 0
Time Frame: day 0 to day 365
Measure: Mean (Standard Deviation); unit: Percentage of patients
Arm/Group | Single Arm Group
Number analyzed (Participants) | 14
Percentage of patients | 0 (0)

3. Secondary Outcome: Plasma C-peptide
Description: Level of plasma C-peptide at 1 year after the first transplant
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Single Arm Group
Number analyzed (Participants) | 14
ng/ml | 1.7 (0.9)

4. Secondary Outcome: HbA1c < 6.5%
Description: The percentage of subjects with HbA1c < 6.5% at 1 year after the first transplant
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Single Arm Group
Number analyzed (Participants) | 14
Percentage of participants | 64.3 (35.7)

5. Secondary Outcome: Percentage of Time Spent in Hypoglycemia (<0.70 mg/L)
Description: percentage of time spent in hypoglycemia derived from CGMS (Continuous Glucose Monitoring System)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Single Arm Group
Number analyzed (Participants) | 14
percentage of time | 11.37 (3.92)

6. Secondary Outcome: Number of Adverse Events
Description: The number of adverse events related to the procedure and to the immunosuppression
Time Frame: 1 year
Measure: Number; unit: number events
Arm/Group | Single Arm Group
Number analyzed (Participants) | 14
number events | 33

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Single Arm Group
Serious Adverse Events (participants affected / at risk) | 12/14
Other Adverse Events (participants affected / at risk) | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Group (N=14)
anemia (Blood and lymphatic system disorders) | 3 (5)
choleperitonitis (Hepatobiliary disorders) | 1 (1)
cholestasis (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (3)
Increase of creatinin (Renal and urinary disorders) | 1 (1)
Increase of SGPT (Hepatobiliary disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 4 (11)
Incarcerated hernia (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
hemocholecyst (Hepatobiliary disorders) | 1 (1)
proteinuria (Renal and urinary disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Group (N=14)
oral ulcerations (Skin and subcutaneous tissue disorders) | 5 (10)
leg edema (Skin and subcutaneous tissue disorders) | 2 (2)
dermatosis (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No